CLINICAL TRIAL: NCT03889249
Title: Alteplase Compared to Tenecteplase in Patients With Acute Ischemic Stroke: QuICR & OPTIMISE Registry Based Pragmatic Randomized Controlled Trial
Brief Title: Alteplase Compared to Tenecteplase in Patients With Acute Ischemic Stroke
Acronym: AcT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Bijoy Menon, Stroke Neurologist, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 2.0 (Sponsor assigned)
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Stroke, Acute; Thromboses, Intracranial
MeSH Terms: conditions — Stroke; Intracranial Thrombosis | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: The proposed trial is a pragmatic, registry linked, prospective, randomized (1:1) controlled, open-label parallel group clinical trial with blinded endpoint assessment of 1600 patients to test if intravenous tenecteplase (0.25 mg/kg body weight, max dose 25 mg) is non-inferior to intravenous alteplase (0.9 mg/kg body weight) in patients with acute ischemic stroke otherwise eligible for intravenous thrombolysis as per standard care.
Who Masked: Outcomes Assessor
Masking Description: 90 day outcomes are assessed in a blinded manner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase (tNK-TPA) (Active Comparator): The intervention group will receive intravenous tenecteplase as a single bolus as per the standard manufacturers' instructions for use. The dose administered will be 0.25 mg/kg body weight (maximum dose 25 mg) over 10-20 seconds as soon as possible after randomization. Tenecteplase has a longer half-life, is more fibrin specific, produces less systemic depletion of circulating fibrinogen, and is more resistant to plasminogen activator inhibitor than alteplase.
  Interventions: Drug: Tenecteplase
- Alteplase ( tPA) (Active Comparator): The control group will receive standard of care dosing of intravenous alteplase (0.9 mg/kg body weight, 10% bolus and 90% infusion as per standard care, maximum dose 90 mg).
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tenecteplase — Stroke Thrombolytic
  Other Names: tNK
  Arms: Tenecteplase (tNK-TPA)
Drug: Alteplase — Stroke Thrombolytic
  Other Names: tPA
  Arms: Alteplase ( tPA)

SUMMARY:
The proposed trial is a pragmatic, registry linked, prospective, randomized (1:1) controlled, open-label parallel group clinical trial with blinded endpoint assessment of 1600 patients to test if intravenous tenecteplase (0.25 mg/kg body weight, max dose 25 mg) is non-inferior to intravenous alteplase (0.9 mg/kg body weight) in patients with acute ischemic stroke otherwise eligible for intravenous thrombolysis as per standard care. All patients will have standard of care medical management on an acute stroke unit. There are no additional trial specific management recommendations. Patients will be followed for approximately 90-120 days.

DETAILED DESCRIPTION:
There are two established therapies for acute ischemic stroke, namely intravenous alteplase and endovascular thrombectomy (EVT). The guiding principles behind these therapies are fast, effective and safe reperfusion of ischemic brain. Patients with acute ischemic stroke presenting within 4.5 hours from symptom onset are administered intravenous alteplase. If there is evidence of large vessel occlusion (LVO), these patients are transferred to the nearest comprehensive stroke center (CSC) for EVT.Physicians, hospitals and health systems are focused on implementing efficient triaging systems and workflow processes to improve speed and efficacy of administration of these life-saving therapies. Although efforts over the years with intravenous alteplase administration has resulted in improvement in efficiency metrics like door to needle time (DTN) and door-in-door-out (DIDO) time, these metrics are still not optimal, and the therapy is underutilized. Physicians continue to have concerns about low early reperfusion rates, increased risk of symptomatic intracerebral hemorrhage and challenges with drug administration (bolus + 60-minute infusion) with intravenous alteplase.

Recent phase II trials have shown that intravenous tenecteplase is potentially safer and may achieve higher early reperfusion rates than alteplase in patients with acute ischemic stroke. Bolus administration makes tenecteplase easier to administer than alteplase (which requires infusion pumps). Transfer of patients from primary stroke centers (PSC) to comprehensive stroke centers (CSCs) is potentially easier without infusion pumps. Moreover, depending on the province, tenecteplase either costs the same, or even less, than alteplase. It is therefore possible that the use of intravenous tenecteplase in patients with acute ischemic stroke otherwise eligible for intravenous alteplase may result in faster administration of thrombolysis and more efficient transport to CSCs, thus saving time, reducing adverse events (intracranial hemorrhage) and potentially improving patient outcomes, while saving the health system costs. For these various reasons, robust evidence that tenecteplase is non-inferior to alteplase as an intravenous thrombolytic agent in patients with acute ischemic stroke will change current clinical practice as it did in patients with myocardial infarction. The proposed trial is therefore a pragmatic, registry linked, prospective, randomized (1:1) controlled, open-label parallel group clinical trial with blinded endpoint assessment of 1600 patients to generate real world evidence whether intravenous tenecteplase (0.25 mg/kg body weight, max dose 25 mg) is non-inferior to intravenous alteplase (0.9 mg/kg body weight) in patients with acute ischemic stroke otherwise eligible for intravenous thrombolysis as per current standard of care.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria is pragmatic and informed by Canadian Best Practices.

* All patients with acute ischemic stroke eligible to receive intravenous alteplase as per standard care will be eligible for enrolment in the proposed trial.
* Patients eligible for endovascular thrombectomy in addition to intravenous thrombolysis are eligible for enrolment.

Exclusion Criteria:

* Contra-indications to intravenous thrombolysis as used by treating physicians as current standard of care apply.
* The benefits of thrombolysis with intravenous alteplase in the pediatric population is unknown. Any patient < 18 years of age may therefore not be enrolled.
* Women with pregnancy known to the investigator by history or examination, without requiring pregnancy testing, may only be enrolled in consultation with an expert stroke physician (either in person or through tele-stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) 0-1 (freedom from disability) | By telephone Follow-up between 90-120 days
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The mRS is a range from 0-6. 0=No symptoms, 1=No significant disability. Able to carry out all usual activities, despite some symptoms 2=Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3=Moderate disability. Requires some help, but able to walk unassisted4=Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5=Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6=Dead

SECONDARY OUTCOMES:
Discharge Destination | 90-120 days after randomization
  Location where the patient is living at 90-120 days from randomization. Locations include home, early supported discharge, rehabilitation facility, long term care, death.
Home Time | 90-120 days after randomization
  Defined as number of days subject spends at home after index stroke event. The home time outcome will be determined through linkage with administrative data to calculate the total time in the first 90 days after index event that a stroke patient is not an inpatient.
Door to needle time | Baseline-Day 1
  Time from when the patient enters the Emergency Room until treatment with either tNK or tPA. Secondary outcome measures described above are all available through the QuICR and OPTIMISE registries and will be collected from those data sources.
Door-in-door-out (DIDO) times at Primary Stroke Centres | Baseline - Day 1
  The amount of time from when the patient enters the Emergency room to the time of discharge from the same hospital is collected. Secondary outcome measures described above are all available through the QuICR and OPTIMISE registries and will be collected from those data sources.
Recanalization | Baseline- After Randomization- Day 1-
  Recanalization status (mTICI score) at first angiographic acquisition in patients taken to the angio-suite for the purpose of administering EVT.Secondary outcome measures described above are all available through the QuICR and OPTIMISE registries and will be collected from those data sources.
Proportion of patients administered EVT | After IV thrombolysis -within the first hour after randomization - baseline-Day 1
  Patients receiving Endovascular Therapy after being treated with either tNK or tPA.Secondary outcome measures described above are all available through the QuICR and OPTIMISE registries and will be collected from those data sources.
Door-to-groin puncture time in patients undergoing EVT | During EVT administration-Baseline- after randomization
  Patients receiving Endovascular Therapy after being treated with either tNK or tPA-treatment time. Secondary outcome measures described above are all available through the QuICR and OPTIMISE registries and will be collected from those data sources.
CT-to-puncture time in patients undergoing EVT | Before EVT administration- baseline- after Randomization- Day 1
  Patients receiving Endovascular Therapy after being treated with either tNK or tPA-treatment time. Secondary outcome measures described above are all available through the QuICR and OPTIMISE registries and will be collected from those data sources.
% patients returning to baseline level of functioning | By telephone Follow-up between 90-120 days
  Patient or surrogate reported return to baseline level of functioning

OTHER OUTCOMES:
Death within 90 days | From Baseline- (Randomization) until Day 90
  Collect if the patient died while in the trial and the cause of death.
Number of Patients Diagnosed with a Symptomatic ICH post-acute stroke treatment by CT/MRI | 24 hours days from Baseline- (Randomization)
  Assess any symptomatic ICH related to the tNK or tPA post treatment. AcT defines symptomatic ICH as intracerebral hemorrhage that in the opinion of the investigator is temporally related to and directly responsible for worsening of the neurological condition. While other factors may contribute to neurological worsening, the hemorrhage should, in the investigator's opinion, be the most important factor if there are multiple factors. Thus, the neurological worsening should not be explained better by any other patient condition such as evolution of infarct, hemodynamic alteration, hypoxia etc.

CONTACTS AND LOCATIONS:
Overall Officials: Bijoy K Menon, MD, Principal Investigator — University of Calgary
Locations (22):
- Canada (22):
  - University of Calgary, Calgary, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta
  - Kelowna General Hospital, Kelowna, B.C.
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Halifax Infirmary Queen Elizabeth II, Halifax, Nova Scotia
  - Hamilton Health Sciences General Hospital, Hamilton, Ontario
  - Kingston Health Science Centre, Kingston, Ontario
  - London Health Sciences, London, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - St. Michaels Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - CHUM -Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Univerisite Laval-Hopital de l'Enfant-Jesus, Québec, Quebec
  - Universite de Sherbrooke, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sujanthan S, Rajkumar G, Dainty KN, Barense M, Lanctot KL, Owen AM, Singh N, Buck BH, Khosravani H, Coutts SB, Almekhlafi M, Appireddy R, Tkach A, Catanese L, Dowlatshahi D, Mandzia J, Pikula A, Williams H, Field TS, Manosalva A, Siddiqui M, Hunter G, Horn M, Bala F, Hill MD, Shamy M, Ganesh A, Sajobi T, Menon BK, Swartz RH; AcT Trial Investigators. Faster Thrombolysis Is Associated With Improved Cognitive Outcomes in Patients With Acute Ischemic Stroke Treated With Alteplase and Tenecteplase: A Substudy of the AcT Trial. Stroke. 2025 Oct;56(10):2858-2865. doi: 10.1161/STROKEAHA.125.051670. Epub 2025 Jul 18. PMID 40677228
- [Derived] Singh N, Bala F, Ademola A, Almekhlafi M, Coutts SB, Deschaintre Y, Khosravani H, Buck BH, Appireddy R, Moreau F, Gubitz G, Tkach A, Catanese L, Dowlatshahi D, Medvedev G, Mandzia J, Pikula A, Shankar JJ, Poppe AY, Williams H, Field TS, Manosalva A, Siddiqui M, Zafar A, Imoukhoude O, Hunter G, Shamy M, Demchuk A, Swartz RH, Hill MD, Sajobi TT, Menon BK, Ganesh A. Safety, Functional Disability, Healthcare Utilization, and Quality-of-Life Outcomes in Elderly Receiving Alteplase and Tenecteplase: A Secondary Analysis From the AcT Trial. Stroke. 2025 May;56(5):1169-1179. doi: 10.1161/STROKEAHA.124.049512. Epub 2025 Mar 24. PMID 40123483
- [Derived] Bala F, Diprose W, Menon BK, Singh N, Khosravani H, Tkach A, Catanese L, Dowlatshahi D, Field TS, Hunter G, Sajobi T, Hill MD, Buck BH, Swartz RH, Almekhlafi MA. Effect of thrombolysis type on the efficacy of aspiration versus stent retriever first line thrombectomy: results from the AcT trial. J Neurointerv Surg. 2025 Jun 1;17(e2):e276-e280. doi: 10.1136/jnis-2024-022268. PMID 39379314
- [Derived] Sajobi TT, Arimoro OI, Ademola A, Singh N, Bala F, Almekhlafi MA, Deschaintre Y, Coutts SB, Thirunavukkarasu S, Khosravani H, Appireddy R, Moreau F, Gubitz GJ, Tkach A, Catanese L, Dowlatshahi D, Medvedev G, Mandzia J, Pikula A, Shankar JS, Williams H, Field TS, Manosalva A, Siddiqui M, Zafar A, Imoukhuede O, Hunter G, Demchuk AM, Mishra SM, Gioia LC, Jalini S, Cayer C, Phillips SJ, Elamin E, Shoamanesh A, Subramaniam S, Kate MP, Jacquin G, Camden MC, Benali F, Alhabli I, Horn M, Stotts G, Hill MD, Gladstone DJ, Poppe AY, Sehgal A, Zhang Q, Lethebe B, Doram C, Shamy M, Kenney C, Buck BH, Swartz RH, Menon BK. Quality of Life After Intravenous Thrombolysis for Acute Ischemic Stroke: Results From the AcT Randomized Controlled Trial. Stroke. 2024 Mar;55(3):524-531. doi: 10.1161/STROKEAHA.123.044690. Epub 2024 Jan 26. PMID 38275116
- [Derived] Kim DJ, Singh N, Catanese L, Yu AYX, Demchuk AM, Lloret-Villas MI, Deschaintre Y, Coutts SB, Khosravani H, Appireddy R, Moreau F, Gubitz G, Tkach A, Dowlatshahi D, Medvedev G, Mandzia J, Pikula A, Shankar J, Williams H, Manosalva H, Siddiqui M, Zafar A, Imoukhuede O, Hunter G, Phillips S, Hill MD, Poppe AY, Ademola A, Shamy M, Bala F, Sajobi TT, Swartz RH, Almekhlafi MA, Menon BK, Field TS. Sex-Based Analysis of Workflow and Outcomes in Acute Ischemic Stroke Patients Treated With Alteplase Versus Tenecteplase. Stroke. 2024 Feb;55(2):288-295. doi: 10.1161/STROKEAHA.123.045320. Epub 2024 Jan 4. PMID 38174568
- [Derived] Singh N, Almekhlafi MA, Bala F, Ademola A, Coutts SB, Deschaintre Y, Khosravani H, Buck B, Appireddy R, Moreau F, Gubitz G, Tkach A, Catanese L, Dowlatshahi D, Medvedev G, Mandzia J, Pikula A, Shankar JJ, Ghrooda E, Poppe AY, Williams H, Field TS, Manosalva A, Siddiqui MM, Zafar A, Imoukhoude O, Hunter G, Shamy M, Demchuk AM, Claggett BL, Hill MD, Sajobi TT, Swartz RH, Menon BK. Effect of Time to Thrombolysis on Clinical Outcomes in Patients With Acute Ischemic Stroke Treated With Tenecteplase Compared to Alteplase: Analysis From the AcT Randomized Controlled Trial. Stroke. 2023 Nov;54(11):2766-2775. doi: 10.1161/STROKEAHA.123.044267. Epub 2023 Oct 6. PMID 37800372
- [Derived] Menon BK, Buck BH, Singh N, Deschaintre Y, Almekhlafi MA, Coutts SB, Thirunavukkarasu S, Khosravani H, Appireddy R, Moreau F, Gubitz G, Tkach A, Catanese L, Dowlatshahi D, Medvedev G, Mandzia J, Pikula A, Shankar J, Williams H, Field TS, Manosalva A, Siddiqui M, Zafar A, Imoukhuede O, Hunter G, Demchuk AM, Mishra S, Gioia LC, Jalini S, Cayer C, Phillips S, Elamin E, Shoamanesh A, Subramaniam S, Kate M, Jacquin G, Camden MC, Benali F, Alhabli I, Bala F, Horn M, Stotts G, Hill MD, Gladstone DJ, Poppe A, Sehgal A, Zhang Q, Lethebe BC, Doram C, Ademola A, Shamy M, Kenney C, Sajobi TT, Swartz RH; AcT Trial Investigators. Intravenous tenecteplase compared with alteplase for acute ischaemic stroke in Canada (AcT): a pragmatic, multicentre, open-label, registry-linked, randomised, controlled, non-inferiority trial. Lancet. 2022 Jul 16;400(10347):161-169. doi: 10.1016/S0140-6736(22)01054-6. Epub 2022 Jun 29. PMID 35779553